CLINICAL TRIAL: NCT00329680
Title: Investigating Nutritional Therapy With EPA, GLA and Antioxidants Role in Sepsis Treatment-INTERSEPT STUDY
Brief Title: The Effects of Eicosapentaenoic Acid (EPA), Gamma-Linolenic Acid (GLA) and Antioxidants in the Treatment of Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fernandes Tavora Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Alessandro Pontes-Arruda Md, MSc, PhD, Fernandes Távora Hospital - CEJPLR - Intensive Care and Nutrition Department
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ILAS-04-ABT
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2009-12-31 (Estimated); Status verified 2009-10

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: Sepsis; Severe Sepsis; Septic Shock; Enteral Nutrition; Antioxidants; EPA; GLA; Nutrition; Intensive Care; ICU
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Eicosapentaenoic Acid; gamma-Linolenic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Experimental arm will receive an enteral diet enriched with EPA, GLA and Antioxidant vitamins
  Interventions: Dietary Supplement: Eicosapentaenoic acid, Gamma-Linolenic Acid and Antioxidant Vitamins
- 2 (Placebo Comparator): This arm will receive an enteral diet considered as a "standard" ICU diet, isocaloric to the control diet but not enhanced with EPA, GLA and antioxidant vitamins
  Interventions: Dietary Supplement: Standard ICU enteral diet, isocaloric to the study diet

INTERVENTIONS:
Dietary Supplement: Eicosapentaenoic acid, Gamma-Linolenic Acid and Antioxidant Vitamins — An enteral diet will be given in accordance with the caloric goal calculated by the Harris-Benedict equation x 1.3. The enteral diet will be provided for a period of 7 days or until death OR start of oral diet OR start of parenteral diet OR discharge from the ICU OR decision from the attending physician/family/patient to no longer participate in this clinical study
  Other Names: Oxepa (Ross Products Division, Abbott Laboratories)
  Arms: 1
Dietary Supplement: Standard ICU enteral diet, isocaloric to the study diet — Patients will receive this diet in a blinded way using the same dose regimen specified previously and used in the study group
  Other Names: Osmolite HiCal/Ensure Pkus HN (Ross Products Division, Abbott Laboratories)
  Arms: 2

SUMMARY:
The scope of this clinical study is to evaluate the possible role of an enteral formulation enriched with EPA, GLA and Antioxidants in patients diagnosed in the early stages of sepsis despite mechanical ventilation requirements, as well as the impact of this diet upon glycemic control and its capacity to prevent the development of sepsis into severe sepsis and septic shock.

DETAILED DESCRIPTION:
The effectiveness of nutritional support in modulating the chain of inflammatory response and in reducing demands of the respiratory system through use of nutritional intervention has received a growing attention, as a result of its capacity to interfere in a variety of biological processes [1]. Nutritional formulations that are low in carbohydrates and rich in lipids may reduce minute-ventilation and ventilatory demand, leading to a reduction of respiratory coefficient and CO2 production [2]. Gadek et al. [3] used a high lipid enteral diet enriched with eicosapentaenoic acid (EPA or fish oil), gamma-linolenic acid (GLA or borage oil) and enhanced levels of antioxidant vitamins in patients with ARDS, demonstrating a significant improvement, not only in the PaO2/FiO2 ratio, but also in several outcomes such as ventilator-free days, ICU-free days and reduced new organ dysfunctions. A recent clinical trial demonstrated that the use of this type of diet may produce better outcomes also in patients with acute lung injury (ALI) [4].

Recent pharmaceutical interventions proposed for sepsis have sought to focus on regulating the chain of pro and anti-inflammatory mediators [5,6], responsible for causing the systemic characteristics of the disease and, consequently, for leading to multiple organ failure. The inflammatory reaction is capable of activate synthesis of lipid mediators, such as prostaglandin E2, which are involved in the complex regulation of the inflammatory process [7].

Many of these inflammatory mediators are metabolites of omega-6 fatty acids, such as linoleic acid and the product of its elongation/desaturation, arachidonic acid [8]. Substitution of Omega-6 fatty acids by fatty acids rich in Omega-3, such as EPA, has proved to be beneficial in modulating the inflammatory processes both in animal models and in humans [9-17].

Interest has also grown around the potential metabolic effects of GLA. This oil is rapidly lengthened to dihomo-gamma-linolenic acid (DGLA) and is incorporated into tissue lipids. DGLA may, amongst other effects, suppress bio-synthesis of leukotrienes, being rapidly metabolized to monoenoic prostaglandins [18]. In addition, although EPA allows the elongation of GLA into DGLA, it tends to prevent its desaturation into arachidonic acid. This mechanism can produce an increase in 1 series prostanoids and a decrease in 2 series eicosanoids.

Research using animal models of sepsis-induced ARDS has shown that a diet low in carbohydrates and rich in EPA and GLA may modulate the production of inflammatory mediators, improving the functional capacity of the lungs. This type of diet is capable of rapidly reducing the phospholipid fatty acid content of arachidonic acid in inflammatory cell membranes [19], even if administered parenterally [20]. In animal models of sepsis, a diet enriched with omega-3 fatty acids has been associated with reduced mortality [21-24].

Moreover, a recent study [25] demonstrated the beneficial effects of an enteral diet enriched with EPA, GLA and elevated level of antioxidant vitamins, in patients with severe sepsis and septic shock requiring mechanical ventilation. In this subpopulation of patients, the use of an enteral formulation enriched with EPA, GLA and Antioxidants is associated with an improvement in oxygenation status, reduced mechanical ventilation time, fewer days in ICU, less new organ dysfunction and also with a 19.4% absolute risk reduction in mortality (NNT=5). Since there is evidence in the literature pointing towards the anti-inflammatory roles not only of EPA and GLA (26), but also of antioxidant vitamins alone (27-29), the differences between both groups may be explained not just by the effects of EPA, GLA or antioxidants, but also by a combination of them. Although this and the previously published trials were designed to investigate the effect of this diet in patients with ARDS, certain differences prove to be particularly relevant. First, the former study examines the effects of such a diet in a population of ARDS patients constituted solely by patients with severe sepsis or septic shock. Moreover, it enrolled patients with a PaO2/FiO2 ratio below 200, rather than below 250, as occurred in the latter study. The heightened gravity of the patients used may have contributed to the greater number of days requiring mechanical ventilation and lower days outside ICU, when compared with previously published results. Finally, this study allows only 6 hours from the moment at which patients fulfilled all entry requirements to effective onset of diet, rather than 24 hours, leading to a significant reduction in time necessary to achieve 75% of BEE x 1.3. Recent studies have shown that time-dependence is a determinant aspect in the treatment of septic patients.

For instance, the PROWESS study [5] showed a significant reduction in the mortality of severe septic patients with a high APACHE II score and who were treated with recombinant human activated protein C (rhAPC) in the first 48 hours after fulfillment of study entry criteria. Nevertheless, the ENHANCE study showed that septic patients who were treated with rhAPC in the first 24 hours after meeting inclusion criteria had lower mortality than those patients who were treated after 24 hours, but within the first 48 hours. The early use was also associated with a lower consumption of hospital resources including mechanical ventilation and the use of vasopressors [30]. Time-dependency was also associated with several other recommendations for the management of septic patients [31].

Another important finding from this recent trial is the number of patients who developed new organ failures not observed at the baseline, considerably lower in the group that received the study diet. This reduction demonstrates a trend towards lower evolution of multiple organ dysfunction in patients fed with EPA+GLA+Antioxidants. If we consider that the development of multiple organ dysfunctions is associated with increasing mortality rates, we can hypothesize this may be a determining factor in reducing the mortality rate [32]. This also suggested that this diet may develop an important role for patients in the early stages of sepsis, by preventing the evolution of the disease to severe sepsis or septic shock.

On the other hand, hyperglycemia and insulin resistance are common in critically ill patients, even when glucose homeostasis has previously been normal. Increased gluconeogenesis, despite abundantly released, is probably central to this disruption of glucoregulation [33,34]. Strict maintenance of normoglycemia with intensive insulin therapy has been shown to reduce intensive care and hospital mortality and morbidity of critically ill adult patients [35].

Supplements or tube feeding using standard nutritional formulations can significantly compromise glycemic control [36-39], very probably due to the rapid and efficient absorption of these liquids. This is specially relevant in those individuals with overt diabetes or stress-related glucose intolerance, such as occurred in septic patients. In such individuals the use of standard nutritional formulations may complicate attempts to achieve and maintain normoglycemia. The answer for this matter may remain in the use of enteral diets high in lipids and low in carbohydrates.

The scope of this clinical study is to evaluate the possible role of an enteral formulation enriched with EPA, GLA and Antioxidants in patients diagnosed in the early stages of sepsis despite pulmonary failure, as well as the impact of this diet upon glycemic control and its capacity to prevent the development of sepsis into severe sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, at the intensive care unit with diagnosis of sepsis and requiring enteral nutrition
* The diagnosis of sepsis follow the criteria previously defined by Bone et al., and modified in accordance with Bernard GR et al
* Included patients MUST start enteral feeding within 12 hours after fulfillment of all inclusion criteria to be considered evaluable
* In addition, patients MUST achieve at least once 75% of BEE (calculated using the Harris-Benedict equation) x 1.3 to be considered evaluable
* Patient septic state and caloric intake will be accessed in a daily basis

Exclusion Criteria:

* Patients with septic shock at the baseline
* Pregnancy or breastfeeding
* Patients under 18 years of age
* Significant limitation of survival prognosis (patients expecting a life survival under 28 days due to a chronic and/or incurable disease such as uncontrolled cancer or other terminal disease)
* Pre-existing chronic renal insufficiency and need of hemodialysis or peritoneal dialysis
* Acute pancreatitis without established origin
* Participation in other clinical trial less than 30 days before inclusion in this trial
* Head trauma with a Glasgow Come Score (GCS) less or equal to 5
* Recent stroke or subarachnoid hemorrhage (less than 3 months)
* Severe immunologic suppression (defined as a leukocyte count bellow 5.000 cells/mm3)
* Infection by the human immunodeficiency virus
* Patients with no indication for enteral feeding or in the imminence of receiving parenteral nutrition
* Patients receiving partial parenteral nutrition in order to achieve caloric goal
* Presence of uncontrolled diarrhea
* Recent gastrointestinal bleeding event
* Patient's, patient's legal representative or physicians decision to exclude patients from this protocol, known hypertriglyceridemia, obesity with BMI over 29.9.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Evolution to more severe forms of the disease | 28-days follow up

SECONDARY OUTCOMES:
28 days all-cause mortality,hyperglycemia, hypoglycemia, mean dose of insulin, use of hospital resources, ICU-free days,creatinine clearance, development of new organ failure,Evolution of the SOFA | 28-days follow up

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Pontes-Arruda, MD, PhD, Principal Investigator — Hospital Fernandes Távora
Locations (12):
- Brazil (12):
  - Hospital Fernandes Távora - Adult Intensive Care Unit, Fortaleza, Ceará
  - Hospital Português - Real Sociedade Portuguesa 16 de Setembro, Salvador, Estado de Bahia
  - Hospital Salvador, Salvador, Estado de Bahia
  - Hospital Santa Luzia, Brasília, Federal District
  - Hospital de Clínicas da Universidade Federal da Paraíba, João Pessoa, Paraíba
  - Clínica São Vicente, Rio de Janeiro, Rio de Janeiro
  - Hospital Pró-Cardíaco, Rio de Janeiro, Rio de Janeiro
  - Associação Beneficente Evangélica de Joinville - Hospital Dona Helena, Joinville, Santa Catarina
  - Centro Hospitalar Unimed, Joinville, Santa Catarina
  - Fundação Faculdade de Medicina de São José Do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital São Paulo-UNIFESP, São Paulo, São Paulo
  - Instituto de Assistência Médica Ao Servidor Público Estadual-Iamspe, São Paulo, São Paulo

REFERENCES:
- See also: Latin American Sepsis Institute Homepage — http://www.sepsisnet.org